CLINICAL TRIAL: NCT06195878
Title: Sleep Apnea in Paralympic Ontario-Resident aThletes With Spinal Cord Injury (SPORTS) Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Julio Furlan, MD, Julio C Furlan, MD, PhD, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-5716
Record Dates: First submitted 2023-12-24; First posted 2024-01-08 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Sleep Apnea; Breathing Disorder During Sleeping; Sleep Disorder; Spinal Cord Injuries; Spine Disease
Keywords: sleep-related breathing disorders; sleep apnea; Spinal Cord Injuries; para-athletes; Spinal Diseases; sports
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Wake Disorders; Spinal Cord Injuries; Spinal Diseases

STUDY DESIGN:
Intervention Model Description: Device: Continuous positive airway pressure (CPAP) therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPAP Therapy (Experimental): Participants who are diagnosed with moderate-to-severe sleep related breathing disorders (SRBDs) will undergo a 4-month trial of Continuous positive airway pressure (CPAP) therapy.
  Interventions: Device: CPAP Therapy

INTERVENTIONS:
Device: CPAP Therapy — Continuous positive airway pressure (CPAP) therapy in the management of moderate-to-severe sleep-related breathing disorders (SRBDs)/sleep apnea.

SUMMARY:
This single arm clinical trial will assess whether continuous positive airway pressure (CPAP) therapy in the management of moderate-to-severe sleep-related breathing disorders (SRBDs) among para-athletes living with cervical/thoracic, complete or incomplete spinal cord injury (SCI) is effective in improving cognitive impairment, in reducing fatigue, depression, anxiety, and overall quality of life. Further, the study will evaluate the effectiveness of CPAP therapy in improving their performance in sports and the perceived risk of injuries.

DETAILED DESCRIPTION:
Untreated moderate-to-severe SRBDs are associated with an increased risk of stroke, heart attack, diabetes, and kidney problems. For para-athletes living with SCI, it can have a major negative impact on their performance when practicing and playing sports.

CPAP therapy is the treatment of choice for moderate-to-severe SRBD (or sleep apnea) in accordance with current good medical practices.

Therefore, the aim of the study is to determine whether CPAP therapy in para-athletes living with SCI who developed moderate-to-severe SRBDs is effective in improving memory, psychosocial implications, social and work participation, and performance in sports.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a cervical or thoracic, complete or incomplete (AIS A to D), chronic (> 6 months) SCI;
* English-speaking adults (18 years of age or older); and
* Play a wheelchair sport at a high-performance level.

Exclusion Criteria:

* A previous history of diagnosis and treatment for sleep apnea;
* Concomitant diseases of the central nervous system and other pre-existing diseases of the central nervous system;
* Current substance misuse;
* History of primary hypersomnia, or secondary hypersomnia of any cause except for SRBDs.
* Conditions that might prevent participants to follow the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Fatigue Severity Scale | Change in Fatigue Severity Scale from baseline to after 4-month period of CPAP therapy
  Self-reported (or administered by an interviewer) scale where participants choose one of seven levels of agreement for each question. Range from 9 (best outcome) to 63 (worst outcome).
Karolinska Sleepiness Scale | Change in Karolinska Sleepiness Scale from baseline to after 4-month period of CPAP therapy
  Measure the level of daytime sleepiness. The scores vary from 1 (normal) to 10 (extremely sleepy).
Medical Outcomes Study Sleep Scale | Change in Medical Outcomes Study Sleep Scale from baseline to after 4-month period of CPAP therapy
  Scores for the sleep disturbance, snoring, respiratory problems, sleep adequacy, and daytime somnolence dimensions range from 0 (normal) to 100.
Depression, Anxiety & Stress Scales- 21 | Change in Depression, Anxiety & Stress Scales- 21 from baseline to after 4-month period of CPAP therapy
  Self-reported (or administered by an interviewer) scale where participants rate questions on depression, anxiety and stress. The DASS-21 scores vary from 0 (normal) to 42 (most severe symptoms of depression, anxiety and stress).
Craig Handicap Assessment and Recording Technique | Change in Craig Handicap Assessment and Recording Technique from baseline to after 4-month period of CPAP therapy
  The CHART assesses capability in 6 domains as follow: physical independence, cognitive independence, mobility, occupation, social integration, and economic self-sufficiency. The scoring for each CHART dimension varies from 0 to 100 points (normal)
SF-36 | Change in SF-36 from baseline to after 4-month period of CPAP therapy
  Patient-reported (or administrated by an interviewer) questionnaire that assesses 8 domains with regards to physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health.
Montreal Cognitive Assessment | Change in Montreal Cognitive Assessment (MoCA) score from baseline to after 4-month period of CPAP therapy
  The Montreal Cognitive Assessment test assess cognitive impairment and scores vary from 0 (worst outcome) to 30 (best outcome).
Recovery-Stress Questionnaire for Athletes (RESTQ-Sport) | aseline (before CPAP therapy) and follow-up assessment (after completion of the 4-month trial of CPAP therapy)
  Assess perceived stress and recovery among athletes. Responses vary from 0 (never) to 6 (always) indicating the frequency of various activities during the past three days and nights. The RESTQ-Sport scores can vary from 0 (best outcome) to 462 (worst outcome).
Acute Recovery and Stress Scale (ARSS) | Change in Acute Recovery and Stress Scale from baseline to after 4-month period of CPAP therapy
  Consists of questions on recovery and stress. The participants are instructed to rate how much each expression applies to them at that moment with responses ranging from 0 (does not apply at all) to 6 (fully applies). The ARSS can vary from 0 (worst outcome) to 192 (best outcome).
Sport Performance Test | Change in Sport Performance Test from baseline to after 4-month period of CPAP therapy
  Sports performance using physiologic tests: Graded Exercise Test (GXT) with VO2 and Sprint Test (Wingate), which will be performed in the physiology laboratory at the Canadian Sport Institute.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Julio Furlan, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Rehab - Lyndhurst Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The UHN REB needs to approve any plan to share data from this study.